CLINICAL TRIAL: NCT04527484
Title: A Single-center, Randomized, Parallel, Open-label , Bioequivalence Study to Compare the Two Formulations of SHR-1314 After Subcutaneous Injection in Healthy Subjects
Brief Title: A Bioequivalence Study to Compare Two Formulations of SHR-1314 After Subcutaneous Injection in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SHR-1314-105
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Bioequivalence

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): SHR-1314 Vial
  Interventions: Drug: SHR-1314
- Group B (Active Comparator): SHR-1314 PFS
  Interventions: Drug: SHR-1314

INTERVENTIONS:
Drug: SHR-1314 — each group subjects will be given different formulations of SHR-1314

SUMMARY:
This study will be a single-center, randomized, parallel, open-label, single dosing bridging study in healthy subjects to evaluate bioequivalence of two formulations of SHR-1314. Subjects will be randomly assigned to the Vials group, the PFS group at a ratio of 1:1

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study related activity is performed. Where relevant, a legal representative will also sign the informed study consent according to local laws and regulations
* Men or women at least 18 years and no more than 45 years of age at time of screening.
* Men with a body weight ≥50 kg or women with a body weight ≥45kg, with BMI range from 18 to 25.
* Subjects with normal physical examination results and with normal laboratory results (blood, chemistry, urine, drug screening, coagulation function test), ECG and X-ray chest test are normal or with certain abnormal without clinical significance.

Exclusion Criteria:

* Presence of significant medical problems, with investigator's judge that not proper to participate clinical study
* History of hypersensitivity to any of study drug constituent
* History or current infection with human immunodeficiency virus (HIV) or hepatitis C; or current hepatitis B infection or syphilis
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years
* History of chronic or recurrent infectious disease, or evidence of active or latent tuberculosis infection.
* Those who have participated in any clinical study for any drug or medical device within 3 months before screening
* Those who have been vaccinated with live attenuated vaccine within 12 weeks prior to screening
* History or evidence of ongoing alcohol or drug abuse, within the last six months before Baseline.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Subjects judged by the investigator as unsuitable for participating in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-last: Area under the serum concentration-time curve from time zero to the last measurable concentration | from Day1 to Day113
  Compare the AUC0-last of 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects
Cmax: Observed maximum serum concentration | from Day1 to Day113
  Compare the Cmax of 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects
AUC0-∞: Area under the serum concentration-time curve from time zero to infinity | from Day1 to Day113
  Compare the AUC0-∞ of 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects

SECONDARY OUTCOMES:
Tmax : Time at which observed maximum concentration occurs | from Day1 to Day113
  Compare the Tmax of 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects
CL/F: Apparent clearance | from Day1 to Day113
  Compare the CL/F of 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects
t1/2: Terminal half-life | from Day1 to Day113
  Compare the t1/2 of 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects
V/F:Apparent volume of distribution | from Day1 to Day113
  Compare the V/F of 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects
Incidence and severity of adverse events (AEs). | from Day1 to Day113
  Compare Incidence and severity of AE at 240mg subcutaneous injection of two specifications of SHR-1314 injection in healthy subjects
Anti-drug Antibodies (ADAs) | from Day1 to Day113
  Incidence of development of Anti-drug Antibodies (ADAs) during the course of the study.

IPD SHARING:
Plan to Share IPD: No